CLINICAL TRIAL: NCT06604910
Title: The Impact of Oral Branched-Chain Amino Acids Under Enhanced Recovery After Surgery on Reducing Postoperative Muscle Loss, Swallowing Difficulties, and Complications After Lower Limb Bone Cancer Curettage for Bone Metastasis
Brief Title: Branched Chained Amino Acid Supplement in Patients Undergoing Lower Limb Bone Cancer Curettage for Bone Metastasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, MD, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202407030RIND
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Muscle Loss
Keywords: nutrition in bone metastases
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: patient undergoing branched chained amino aicd
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCAA (Experimental): patients undergoing branched chained amino acid
  Interventions: Dietary Supplement: branched chained amino acid
- patients undergoing no BCAA (No Intervention): patients undergoing no branched chained amino acid

INTERVENTIONS:
Dietary Supplement: branched chained amino acid — patients undergoing branched chained amino acid
  Arms: BCAA

SUMMARY:
Postoperative muscle loss is common in patients with bone metastases undergoing lower limb bone cancer curettage, affecting both limb skeletal muscles and potentially swallowing-related muscles. Rectus femoris thickness, measured via ultrasound on postoperative day seven, is used to assess this loss. Branched-chain amino acids (BCAAs) are important for muscle protein synthesis, but little research exists on whether postoperative oral BCAA supplementation can reduce muscle loss, swallowing function deterioration, and short-term complications. This study investigates if BCAA supplementation from postoperative day one to day 30 can reduce muscle loss (primary endpoint: rectus femoris thickness on day seven) and mitigate swallowing function decline, pharyngeal muscle contraction loss, and complications within three months post-surgery.

DETAILED DESCRIPTION:
Postoperative muscle loss is common in patients with bone metastases undergoing lower limb bone cancer curettage, affecting both limb skeletal and swallowing-related muscles, with rectus femoris thickness measured via ultrasound on postoperative day seven. Branched-chain amino acids (BCAAs) are crucial for muscle protein synthesis, but limited research exists on whether postoperative oral BCAA supplementation can reduce muscle loss, swallowing function deterioration, and short-term complications within three months. This study aims to determine if BCAA administration from postoperative day one to day 30 can reduce muscle loss, with rectus femoris thickness on day seven as the primary endpoint, while also exploring the effect on swallowing function, pharyngeal muscle strength, and complication rates. It will target patients with lower limb bone metastases from breast, lung, and prostate cancers, excluding those with high mortality risk or metastases in other regions. In a one-year randomized controlled trial, 40 patients will be assigned to receive either 3160 mg of daily BCAA for 30 days or no supplementation. Primary outcomes include rectus femoris muscle thickness and swallowing muscle strength assessed by high-resolution manometry, with postoperative complications followed for three months. The expected result is that the BCAA group will experience less muscle loss, greater rectus femoris thickness, reduced swallowing muscle decline, and fewer complications. This study aims to improve care quality, promote recovery, and support sustainable health goals.

ELIGIBILITY:
Inclusion Criteria:

* I) The patient has a femoral metastasis and is expected to undergo bone tumor curettage and joint replacement surgery, or the patient has a femoral metastasis and is expected to undergo bone tumor curettage and internal fixation surgery; II) Age between 20 and 80 years; III) Able to take care of themselves independently (Karnofsky Performance Status ≥ 70%, which measures a patient's ability to perform daily activities, with a total score of 100 points. A higher score indicates better self-care ability, and a score of 70 or above indicates the ability to live independently but not to work or perform normal daily activities); IV) Patients have all signed a written informed consent.

Exclusion Criteria:

* I) Patients expected to undergo bone tumor curettage and mega prosthesis replacement; II) Patients requiring surgery on both upper and lower limbs; III) Patients requiring surgery on both lower limbs; IV) Patients with simultaneous spinal metastasis; V) Patients likely to undergo a second surgery within 30 days; VI) Patients with metastasis in other locations or a history of metastasis with prior surgeries; VII) Patients with neuromuscular diseases, such as stroke or Parkinson's disease; VIII) Exclusion of patients with other diseases and complications, such as those with concurrent gastric cancer or post-gastrectomy patients requiring additional surgeries due to complications or unstable conditions, patients with New York Heart Association Functional Classification ≥ Class 2 heart disease and thrombotic conditions, patients with Hugh-Jones Classification ≥ Grade 4 lung disease, or those currently receiving insulin therapy; IX) Patients allergic to eggs, soy, or thiamine; X) Patients who are already supplementing BCAAs; XI) Patients with psychiatric disorders that may affect their ability to provide informed consent or comply with the study protocol; XII) If postoperative pathology reveals a diagnosis other than the originally identified cancer metastasis, the case will be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
muscle loss | postoperative one month
  muscle thickness measurement

IPD SHARING:
Plan to Share IPD: No
due ethical issue